CLINICAL TRIAL: NCT04671082
Title: A Phase 3, 14-Day, Double-blind, Randomized, Placebo-Controlled, Multicenter Study of the Efficacy and Safety of Tolperisone in Subjects With Pain Due to Acute Back Muscle Spasm
Brief Title: Efficacy and Safety of Tolperisone in Subjects With Pain Due to Acute Back Muscle Spasm
Acronym: RESUME-1
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Neurana Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CLN-301; RESUME-1 (Other: Neurana Pharmaceuticals)
Record Dates: First submitted 2020-12-10; First posted 2020-12-17 (Actual); Last update posted 2022-03-22 (Actual); Status verified 2022-03

CONDITIONS: Back Muscle Spasm; Back Pain; Back Strain; Back Spasm Upper; Muscle Spasm; Acute Pain
MeSH Terms: conditions — Back Pain; Spasm; Acute Pain | interventions — Tolperisone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Tolperisone 50 mg (Experimental): Tolperisone 50 mg
  Interventions: Drug: Tolperisone Hydrochloride
- Tolpersione 100 mg (Experimental): Tolperisone 100 mg
  Interventions: Drug: Tolperisone Hydrochloride
- Tolperisone 200 mg (Experimental): Tolperisone 200 mg
  Interventions: Drug: Tolperisone Hydrochloride
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Tolperisone Hydrochloride — TID
  Other Names: Tolperisone
  Arms: Tolperisone 200 mg; Tolperisone 50 mg; Tolpersione 100 mg
Drug: Placebo — TID
  Arms: Placebo

SUMMARY:
This is a double-blind, randomized, placebo-controlled, multicenter study of the efficacy and safety of tolperisone (a non-opioid) or placebo administered in subjects with pain due to acute back muscle spasm.

ELIGIBILITY:
Inclusion Criteria:

* Ambulatory
* Current acute back pain due to acute muscle spasm starting within 7 days prior to study entry (Day 1) and at least 8 weeks following resolution of the last episode of acute back pain.
* Willingness to discontinue all previous or ongoing treatment of pain or muscle spasm on study entry at Day 1 through the end of treatment including medication, acupuncture, chiropractic adjustment, massage, transcutaneous electrical nerve stimulation [TENS], or physiotherapy.
* Pain must be localized from the neck (C-3 or lower) to the inferior gluteal folds and spasm assessed during the Screening physical examination.
* Body mass index range between 18 and 35 kg/m², inclusive.

Exclusion Criteria:

* Presence of acute or chronic back pain for the previous 8 days or longer, where back pain is present on more days than not.
* Presence of neurogenic pain in the back, neck, upper or lower extremities, including pain from (or suspected from) nerve root compression or injury (radicular pain or "pinched nerve") or neuropathic pain. Evidence of these types of exclusionary pain includes radiation of pain that radiates beyond the back, chronic pain, and pain associated with abnormal sensation or loss of sensation in the back or extremities.
* Presence of pain anywhere other than the target back pain that is bothersome, interferes with activity, or for which pain relief is taken.
* History of any neck, back, or pelvic surgery.
* History within the previous 3 years of: spinal fracture or spinal infection; inflammatory arthritis; degenerative spine disease; or any other back or spine condition that may reasonably contribute to current back pain.
* Subjects who test positive for alcohol by breathalyzer test or have a positive urine drug screen for drugs of abuse (e.g. amphetamines, methamphetamines, barbiturates, benzodiazepines, cocaine, cannabinoids, oxycodone, opiates), including cannabis even where legal, at Screening.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 1004 (Actual)
Dates: Start 2020-12-15 (Actual); Primary Completion 2021-12-13 (Actual); Study Completion 2022-03-21 (Actual)

PRIMARY OUTCOMES:
Numerical rating scale (NRS) | Day 1 to Day 14
  Numerical rating scale (NRS), a 0-10 scale, from no pain to worst possible pain - Subject-rated pain "right now" due to acute back spasm.

CONTACTS AND LOCATIONS:
Locations (55):
- United States (55):
  - Clinical Research Institute of Arizona, LLC, Surprise, Arizona
  - Applied Research Center of Arkansas, Little Rock, Arkansas
  - Alliance Research Institute, Canoga Park, California
  - Long Beach Clinical Trials Services, Inc, Long Beach, California
  - Northern California Research, Sacramento, California
  - Collaborative Neuroscience Research, LLC, Torrance, California
  - Lynn Institute of Denver, Aurora, Colorado
  - Emerson Clinical Research Institute, Washington D.C., District of Columbia
  - Multi-Specialty Research Associates, Inc., Lake City, Florida
  - LCC Medical Research Institute, LLC, Miami, Florida
  - Savin Medical Group, Miami Lakes, Florida
  - Accel Research Sites, Orange City, Florida
  - Combined Research Orlando, Orlando, Florida
  - iResearch Atlanta, Decatur, Georgia
  - Georgia Clinical Research LLC, Lawrenceville, Georgia
  - IMA Clinical Research, PC, Chicago, Illinois
  - Evanston Premier Healthcare Research LLC, Evanston, Illinois
  - Investigators Research Group, Brownsburg, Indiana
  - Professional Research Network of Kansas, LLC, Wichita, Kansas
  - Research Integrity, LLC, Owensboro, Kentucky
  - DelRicht Research, New Orleans, Louisiana
  - DelRicht Research, Prairieville, Louisiana
  - Michigan Head Pain and Neurological Institute, Ann Arbor, Michigan
  - Onyx Clinical Research, Rochester Hills, Michigan
  - Quinn Healthcare/SKYCRNG, Ridgeland, Mississippi
  - IMA Clinical Research, St Louis, Missouri
  - Pioneer Clinical Research, LLC, Bellevue, Nebraska
  - Skyline Medical Center, PC, Elkhorn, Nebraska
  - Jubilee Clinical Research, Inc., Las Vegas, Nevada
  - Albuquerque Clinical Trials, Inc., Albuquerque, New Mexico
  - Integrative Clinical Trials, LLC, Brooklyn, New York
  - Drug Trials America, Hartsdale, New York
  - Manhattan Behavioral Medicine PLLC, New York, New York
  - Advanced Research Solutions, LLC, Staten Island, New York
  - Upstate ClinicalResearch Associates LLC, Williamsville, New York
  - Carolina Research Center, Inc., Shelby, North Carolina
  - Progressive Medicine of the Triad, LLC, Winston-Salem, North Carolina
  - Hometown Urgent Care and Research, Cincinnati, Ohio
  - Hometown Urgent Care and Research, Columbus, Ohio
  - Hometown Urgent Care and Research, Dayton, Ohio
  - Onyx Clinical Research, Youngstown, Ohio
  - Today Clinical Research, Oklahoma City, Oklahoma
  - DelRicht Research, Tulsa, Oklahoma
  - Frontier Clinical Research, LLC, Smithfield, Pennsylvania
  - PCPMG Clinical Research Unit, LLC, Anderson, South Carolina
  - New Phase Research & Development, LLC, Knoxville, Tennessee
  - Central Texas Clinical Research, Austin, Texas
  - Premier Family Physicians, Austin, Texas
  - ClinRx Research Joseph INC, Carrollton, Texas
  - Centex Studies, Inc., Houston, Texas
  - R & H Clinical Research, Katy, Texas
  - Village Health Partners, Plano, Texas
  - Sun Research Institute, San Antonio, Texas
  - Spectrum Medical, Inc., Danville, Virginia
  - Health Research of Hampton Roads, Inc., Newport News, Virginia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Vaughan SA, Torres K, Kaye R. RESUME-1: a Phase III study of tolperisone in the treatment of painful, acute muscle spasms of the back. Pain Manag. 2022 Jan;12(1):25-33. doi: 10.2217/pmt-2021-0041. Epub 2021 Jul 1. PMID 34192885